CLINICAL TRIAL: NCT03539471
Title: Current Trend of Epidemiology of Psychiatric Emergency and the Stress of Duty Psychiatric Resident
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201708099RIND
Record Dates: First submitted 2018-05-17; First posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2017-10

CONDITIONS: Emergent Psychiatric, Consultation, Residentship

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- psychiatric resident in NTUH
  Interventions: Diagnostic Test: interview, Tridimensional Personality Questionnaire

INTERVENTIONS:
Diagnostic Test: interview, Tridimensional Personality Questionnaire — interview of the residents about 15-20 minutes, then use Tridimensional Personality Questionnaire

SUMMARY:
Agitation, paranoia, and suicide risk of the psychiatric patients made them difficult to be managed when they visited medical emergency services. The prolonged waiting time at medical emergency services and the stigmatization of psychiatric medicine also made the psychiatric emergency services full of challenges. However, in recent years, the random killings, celebrity suicide and other major social events attracted much attention to the emergency psychiatry.

Following the establishment of the National Health Insurance, the law of mandatory admission, and the prevalence change of all psychiatric diseases, we are now dealing with totally different types of emergent psychiatric conditions, i.e., depression and suicide. However, the real epidemiological data need to be updated. Psychiatric emergency is one of the entrances of the psychiatric network. A comprehensive review of the psychiatric emergency would be needed for the base of further research.

This study is aimed to investigate the prevalence of psychiatric diagnosis of patients who came to Emergency Department of National Taiwan University Hospital and needed a psychiatric consultation. The epidemiological data will be compared to those collected 30 years ago in the same hospital to examine the 30-year trend. On the other hand, the visiting time and the staying time will be analyzed. The stress of on-duty and the contributing factors will be assessed by a 2-hour in-depth interview with psychiatric residents.

ELIGIBILITY:
Inclusion Criteria:

* Psychiatric resident in NTUH

Exclusion Criteria:

* Major psychiatric illness

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: NTUH has 4 psychiatric residents each year, from R1 to R4.
Sampling Method: Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative Research | until 2018/11/1
  for 16 residents, interview data

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan